CLINICAL TRIAL: NCT03774979
Title: A Phase I, Open-label Trial to Investigate the Safety, Tolerability, Pharmacokinetics, Biological and Clinical Activity of SHR-1701 in Subjects With Metastatic or Locally Advanced Solid Tumors With Expansion to Selected Indications
Brief Title: SHR-1701 in Subjects With Metastatic or Locally Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1701-I-102
Record Dates: First submitted 2018-12-10; First posted 2018-12-13 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-07

CONDITIONS: Solid Tumor
Keywords: SHR-1701; Solid tumor; Metastatic or locally advanced solid tumors
MeSH Terms: conditions — Neoplasm Metastasis | interventions — SHR-1701

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1701 (Experimental): intravenous infusion
  Interventions: Drug: SHR-1701

INTERVENTIONS:
Drug: SHR-1701 — Subjects will receive an intravenous infusion of SHR-1701 in a pre-set dose escalation until confirmed progression, unaccepted toxicity, or any criterion for withdrawal from the trial.

SUMMARY:
The main purpose of this study is to assess the safety and tolerability of SHR-1701 at different dose levels. Study consists of dose-escalation part and an expansion part in subjects with metastatic or locally advanced solid tumors.

DETAILED DESCRIPTION:
This is a Phase I, open-label, multiple-ascending dose trial. Study consists of dose-escalation part in subjects with metastatic or locally advanced solid tumors, and expansion part with selected indications.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide signed informed consent form, and able to comply with all procedures.
* Histologically or cytologically proven metastatic or locally advanced solid tumors.
* Male or female subjects aged 18-75 years.
* Life expectancy >= 12 weeks as judged by the Investigator.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 at trial entry.
* Disease must be measurable with at least 1 uni dimensional measurable lesion by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* Adequate hematological, hepatic and renal function as defined in the protocol

Other protocol-defined inclusion criteria could apply.

Exclusion Criteria:

* Prior therapy with an anti-PD1, anti-PD-L1, anti-CTLA-4 or a TGFb inhibitor.
* Anticancer treatment within 28 days before the first dose of study drug.
* Major surgery within 28 days before start of trial treatment.
* Systemic therapy with immunosuppressive agents within 7 days prior to the first dose of study drug; or use any investigational drug within 28 days before the start of trial treatment.
* With any active autoimmune disease or history of autoimmune disease.
* With active central nervous system (CNS) metastases causing clinical symptoms or requiring therapeutic intervention.
* Clinically significant cardiovascular and cerebrovascular diseases
* History of immunodeficiency including seropositive for human immunodeficiency virus (HIV), or other acquired or congenital immunedeficient disease, or any active systemic viral infection requiring therapy.
* Previous malignant disease (other than the target malignancy to be investigated in the trial) within the last 2 years. Subjects with history of cervical carcinoma in situ, superficial or non-invasive bladder cancer or basal cell or squamous cell cancer in situ previously treated with curative intent are NOT excluded.
* Receipt of any organ transplantation, including allogeneic stem-cell transplantation

Other protocol-defined exclusion criteria could apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Dose escalation part： Safety and tolerability of SHR-1701 in advanced malignancies. | Up to 3/4 weeks.
  Number of Subjects who occurs dose-limiting toxicity (DLTs).
Clinical expansion Part: Objective Response Rate（ORR） | Up to 6 weeks
  ORR is define as the percentage of participants in the analysis population who havea Complete Response(CR:Disappearance of all target lesions)or a Partial Response(PR :30% decrease in the sum of diameter of target lesions) per RECIST 1.1.

SECONDARY OUTCOMES:
Clinical expansion Part: Safety of SHR-1701 | Up to 4 weeks after last treatment
  Number of subjects who occurs treatment-related Adverse Events(AEs）
Clinical expansion Part: Disease Control Rate(DCR) per RECIST1.1 | Up to 6 weeks
  DCR is define as the percentage of participants in the analysis population who have a CR,PR or SD per RECIST 1.1.
Clinical expansion Part: Duration of Response （DOR）per RECIST1.1 | Up to 6 weeks
  DOR is define as the time from first documented evidence of CR or PR until disease progression per RECIST 1.1
Clinical expansion Part:Progression-free survival(PFS) per RECIST1.1 | 12months (anticipated)
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Jifeng Feng, MD, Principal Investigator — Jiangsu Cancer Institute & Hospital
Locations (16):
- China (16):
  - Anhui Chest Hospital-Departmen of Tumor Radiotherapy, Hefei, Anhui
  - The First Affiliated Hospital of Guangzhou University of Chinese Medicine-Cancer Center, Guangzhou, Guangzhou
  - Xinxiang Central Hospital-Department of Respiratory Physicians, Xinxiang, Henan
  - The First Affiliated Hospital of Zhengzhou University-Department of Medical Oncology, Zhengzhou, Henan
  - Cancer Hospital of Hunan Province, Changsha, Hunan
  - Hunan Cancer Hospital-Gynecologic Oncology, Changsha, Hunan
  - Jangsu Cancer Hospital, Nanjing, Jiangsu
  - The First Rffiurted Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of China Medical University-Department of Oncology, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Sir Run Run Shaw Hospital, Zhejiang University, School of Medicine, Hangzhou, Zhejiang
  - Beijing Chest Hospital,Capital Medical University-Integrated Department, Beijing
  - Tumor Hospital of the Chinese Academy of Medical Sciences, Beijing
  - ChongQing Cancer Hospital-gynecologic oncology, Chongqing
  - Chongqing Cancer Hospital, Chongqing

IPD SHARING:
Plan to Share IPD: No